CLINICAL TRIAL: NCT00414388
Title: Phase I/II Study to Evaluate the Ability of Sorafenib in Overcoming Resistance to Systemic Chemotherapy in Androgen-independent Prostate Cancer (AIPC)
Brief Title: Sorafenib to Overcome Resistance to Systemic Chemotherapy in Androgen-independent Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oncology Specialists, S.C. (Other)
Responsible Party: Principal Investigator, Dr. Sigrun Hallmeyer, Director of Research, Oncology Specialists, S.C.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0603
Record Dates: First submitted 2006-12-19; First posted 2006-12-21 (Estimated); Results first posted 2014-04-07 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-02

CONDITIONS: Prostate Cancer
Keywords: AIPC
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single agent Sorafenib (Experimental): Oral Single agent Sorafenib 400mg twice daily
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Sorafenib — 400mg twice daily
  Other Names: Nexavar

SUMMARY:
The primary objective of this study is to evaluate the safety of combining Sorafenib and chemotherapy (mitoxantrone or docetaxel) in patients with AIPC.

DETAILED DESCRIPTION:
Patients who have AIPC and are progressing despite systemic chemotherapy will be offered participation in this study. Patients who relapse or progress shortly (within 12 weeks) after discontinuation of chemotherapy with either docetaxel/prednisone or mitoxantrone/prednisone will also be offered participation in this trial. Enrolled patients will receive sorafenib as per protocol define dose. Sorafenib will be administered in combination with the last chemotherapy utilized. If there is no disease progression after 6 cycles, chemotherapy will be stopped and Sorafenib may continue until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0, 1, or 2.
* Patients with a known diagnosis of prostate cancer regardless of their Gleason grade.
* Patients have AIPC.
* Adequate bone marrow, liver and renal function as assessed by:
* Hemoglobin > 9.0 g/dl
* absolute neutrophil count (ANC) > 1,000/mm3
* Platelet count > 75,000/mm3
* Total bilirubin < 1.5 x upper limit of normal (ULN)
* Alanine transaminase (ALT) and aspartate aminotransferase (AST) < 2.5 x the ULN (< 5 x ULN for patients with liver involvement). international normalized ratio (INR) < 1.5 or a Prothrombin time (PT)/partial thromboplastin time (PTT) within normal limits. Patients receiving anti-coagulation treatment with an agent such as warfarin or heparin may be allowed to participate.
* Creatinine < 1.5 x ULN
* Transfusions and the use of growth factors (for red and white cells) are allowed
* Patients must have received either docetaxel or mitoxantrone as the chemotherapy regimen
* Ability to understand and willingness to sign a written informed consent. A signed informed consent must be obtained prior to any study specific procedures.
* Patients must have progressed while receiving systemic chemotherapy for AIPC. Patients could have progressed within 12 weeks of their last systemic chemotherapy administration. The definition of progression is defined as follows:

  * 1-For patients who are receiving systemic chemotherapy (one criteria is sufficient):
  * Increase in prostate-specific antigen (PSA) by 25% or more than the previous value. This should be repeated within 3 weeks (while patient is off chemotherapy) to confirm that the PSA did not decrease.
  * For patients with visceral disease, radiographic evidence of progression by standard Response Evaluation Criteria in Solid Tumors (RECIST) criteria (regardless of the PSA value).
  * For patients with bone only disease, progression on a whole body bone scan (2 or more new lesions) is sufficient to fulfill the definition of progressive disease, regardless of PSA value or the visceral disease status.
  * 2-For patients who have received chemotherapy previously (Both criteria are needed):
  * Not more than 12 weeks have elapsed since last chemotherapy administration
  * Either biochemical progression (25% increase in PSA that is confirmed with a repeat analysis within 3 weeks), OR radiographic progression (RECIST criteria for visceral disease patients OR 2 or more lesions on a whole body bone scan)

Exclusion Criteria:

* Cardiac disease: Congestive heart failure > class II New York Heart Association 9NYHA). Patients must not have unstable angina or new onset angina or myocardial infarction within the past 6 months.
* Known brain metastasis. Patients with neurological symptoms must undergo a CT scan or MRI of brain to exclude brain metastasis.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy. Patients with history of chronic and well controlled atrial fibrillation are allowed. Beta-blockers, calcium channel blockers, or digoxin are not considered anti-arrhythmics.
* Uncontrolled hypertension defined as systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management.
* Sorafenib is contraindicated in patients with known severe hypersensitivity to sorafenib or any of the excipients.
* Known human immunodeficiency virus (HIV) infection or chronic Hepatitis B or C.
* Active clinically serious infection > Common Toxicity Criteria for Adverse Effects (CTCAE) Grade 2.
* Thrombolic or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months.
* Pulmonary hemorrhage/bleeding event > CTCAE Grade 2 within 4 weeks of first dose of study drug.
* Any other hemorrhage/bleeding event > CTCAE Grade 3 within 4 weeks of first dose of study drug.
* Serious non-healing wound, ulcer, or bone fracture.
* Evidence or history of bleeding diathesis or uncontrolled coagulopathy.
* Major surgery, open biopsy or significant traumatic injury within 4 weeks of first study drug.
* Use of St. John's Wort or rifampin (rifampicin).
* Known or suspected allergy to sorafenib or any agent given in the course of this trial.
* Any condition that impairs patient's ability to swallow whole pills.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-12; Primary Completion 2011-09 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chadi Nabhan, MD, Principal Investigator — Oncology Specialists, SC
Locations (2):
- United States (2):
  - Onocology Specialists, S.C, Niles, Illinois
  - Oncology Specialists, S.C, Park Ridge, Illinois

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was from our clinic population.
Pre-assignment Details: Eligible patients were those who progressed while receiving chemotherapy (docetaxel or mitoxantrone)or within 12 weeks of stopping chemo.
Groups:
- Single Agent Sorafenib: Eligible patients were continued on the same chemotherapeutic regimen they had progressed on prior on entry into the study (docetaxel or mitoxantrone) with the addition of Sorafenib at 400mg twice daily. Docetaxel was given at 75 mg/m^2 and mitoxantrone was given at 12 mg/m^2, both once every 21 days and both combined with prednisone at 5mg twice daily. A maximum of 6 cycles of sorafenib plus chemotherapy were allowed. Patients without objective disease progression after combination therapy was complete were allowed to receive sorafenib monotherapy until disease progression.
Period: Overall Study
Arm/Group | Single Agent Sorafenib
Started | 22
Completed | 21
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Recruitment was from our clinic population. Eligible patients were those who progressed while receiving chemotherapy (docetaxel or mitoxantrone)or within 12 weeks of stopping chemo
Arm/Group | Single Agent Sorafenib
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 22
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Needing a Dose Reduction.
Description: The actual percentage was determined by taking the number of patients requiring a dose reduction divided by the total number of patients multiplied by100%
Time Frame: participants were followed for an average of 25 months
Population: 15 patients required dose reductions.
Measure: Number; unit: percentage of participants
Arm/Group | Single Agent Sorafenib
Number analyzed (Participants) | 21
percentage of participants | 71 [0 to 100]

2. Secondary Outcome: Overall Clinical Benefit (OCB)of This Combination as Calculated by the Sum of Complete Response (CR), Partial Response (PR), and Stable Disease (SD).
Description: Assessment of response was done per Response Evaluation Criteria in Solid Tumors (RECIST) criteria as outlined in the protocol. Complete Response (CR) defined as disappearance of all measurable lesions. Partial Response (PR) more than 30% decrease in the sum of longest diameter of measurable lesions compared to baseline. Stable Disease (SD) lesions should have no sufficient decrease for PR any sufficient increase to meet criteria for PD. Progressive Disease (PD) more than 20% increase in the sum of longest diameter of measurable lesions compared to baseline, and/or evidence of new lesions on imaging studies or the appearance of 2 or more new bony lesions. For patient with measurable disease,prostate-specific antigen (PSA), progression in the absence of measurable disease progression will not be considered progressive disease. Overall Clinical Benefit (OCB) (CR + PR+ SD)/#participants.
Time Frame: 3-10 months
Measure: Number; unit: percentage of patients
Arm/Group | Single Agent Sorafenib
Number analyzed (Participants) | 21
percentage of patients | 76 [0 to 100]

3. Secondary Outcome: PSA -Biochemical Response
Description: PSA Biochemical Response = PSA complete response + PSA partial response. A PSA complete response is defined as a non-detectable PSA (<4 ng/dl). A PSA partial response is defined as a PSA that decreases by greater than or equal to 50%.
Time Frame: 1-10 months
Measure: Number; unit: percentage of participants
Groups:
- Sorafenib: Eligible patients were continued on the same chemotherapeutic regimen they had progressed on prior on entry into the study (Docetaxel or Mitoxantrone) with the addition of Sorafenib at 400mg twice daily. Docetaxel was given at 75 mg/m2 and Mitoxantrone was given at 12 mg/m2, both once every 21 days and both combined with Prednisone at 5mg twice daily. A maximum of 6 cycles of Sorafenib plus chemotherapy were allowed. Patients without objective disease progression after combination therapy was complete were allowed to receive Sorafenib monotherapy until disease progression.
Arm/Group | Sorafenib
Number analyzed (Participants) | 21
percentage of participants | 45

ADVERSE EVENTS:
Arm/Group | Single Agent Sorafenib
Serious Adverse Events (participants affected / at risk) | 12/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Agent Sorafenib (N=22)
urinary retention (Renal and urinary disorders) | 2
Anemia (Blood and lymphatic system disorders) | 1
Hypoglycemia (General disorders) | 1
constipation (Gastrointestinal disorders) | 2
Back Pain (General disorders) | 1
Electrolyte imbalance (Blood and lymphatic system disorders) | 1
Fatigue (General disorders) | 1
Dehydration (Gastrointestinal disorders) | 1
Adominal Pain (General disorders) | 2
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2
Urinary Tract Infection (Renal and urinary disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
C-diff (Gastrointestinal disorders) | 1
Neutropenic Fever (Blood and lymphatic system disorders) | 1
Diverticular Bleed (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single Agent Sorafenib (N=22)
Fatigue (General disorders) | 16
hand/foot syndrome (Skin and subcutaneous tissue disorders) | 10
Hypoglycemia (General disorders) | 2
Hyperglycemia (General disorders) | 10
Leukopenia (Blood and lymphatic system disorders) | 14
Neutropenia (Blood and lymphatic system disorders) | 9
Thrombocytopenia (Blood and lymphatic system disorders) | 17
Anemia (Blood and lymphatic system disorders) | 17
Lymphopenia (Blood and lymphatic system disorders) | 19
Hypocalcemia (Blood and lymphatic system disorders) | 11
Alopecia (General disorders) | 12
Anorexia (Gastrointestinal disorders) | 15
Albumin decreased (Gastrointestinal disorders) | 15
AST increased (Gastrointestinal disorders) | 6
Alkaline Phosphatase Increased (Gastrointestinal disorders) | 11
Anxiety (Psychiatric disorders) | 4
Arthralgia (Nervous system disorders) | 3
Atrial Fibrillation (Cardiac disorders) | 2
Bruises Easily (Blood and lymphatic system disorders) | 8
Bilirubin Increased (Renal and urinary disorders) | 3
Back Pain (General disorders) | 2
Chills (General disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Concentration Difficulty (General disorders) | 4
Constipation (Gastrointestinal disorders) | 8
Creatinine Increased (Renal and urinary disorders) | 3
Chest pain non cardiac (Musculoskeletal and connective tissue disorders) | 3
Dehydration (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 18
Dizziness (General disorders) | 5
Depression (Psychiatric disorders) | 5
Dyspnea on Exertion (Respiratory, thoracic and mediastinal disorders) | 3
Ear Pain (Ear and labyrinth disorders) | 3
Eyes dry (Eye disorders) | 3
Edema (General disorders) | 4
Eyes tearing (Eye disorders) | 3
Fall (General disorders) | 2
Fever (General disorders) | 4
Foot pain (General disorders) | 2
Facial swelling (General disorders) | 2
Globulin decreased (Gastrointestinal disorders) | 6
Gynecomastia (Reproductive system and breast disorders) | 3
Hard of hearing (Ear and labyrinth disorders) | 3
Hypotension (General disorders) | 2
Hypokalemia (Gastrointestinal disorders) | 8
Headache (General disorders) | 7
Heartburn (Gastrointestinal disorders) | 2
Hypertension (General disorders) | 2
Hyponatremia (Gastrointestinal disorders) | 8
Hot flashes (Reproductive system and breast disorders) | 2
Hyperkalemia (Gastrointestinal disorders) | 4
Itching (Skin and subcutaneous tissue disorders) | 5
Insomnia (General disorders) | 3
Jaw Pain (Musculoskeletal and connective tissue disorders) | 5
Libido decreased (Reproductive system and breast disorders) | 3
Mouth Dry (Gastrointestinal disorders) | 11
Mouth Sores (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 8
Neuropathy (General disorders) | 14
Nail changes (Skin and subcutaneous tissue disorders) | 7
Protein Decreased (Gastrointestinal disorders) | 14
Pain (General disorders) | 7
Pneumonia (Infections and infestations) | 3
Rash (Skin and subcutaneous tissue disorders) | 15
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 4
Skin peeling (Skin and subcutaneous tissue disorders) | 2
Sweats (General disorders) | 3
Stomatitis (Gastrointestinal disorders) | 3
Tachycardia (Cardiac disorders) | 9
Taste Changes (Gastrointestinal disorders) | 7
Throat sore (Gastrointestinal disorders) | 9
Urinary retention (Renal and urinary disorders) | 2
Ulcer pressure (Skin and subcutaneous tissue disorders) | 3
Urination Problems (Renal and urinary disorders) | 3
Vomiting (Gastrointestinal disorders) | 2
Vision Problems (Eye disorders) | 4
Weight decreased (General disorders) | 8
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes